CLINICAL TRIAL: NCT05848180
Title: Effect Of Ankle Proprioceptive Training On Balance And Risk Of Fall In Patients With Diabetic Peripheral Neuropathy
Brief Title: Ankle Proprioceptive Training In Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/Letter-014124
Record Dates: First submitted 2023-04-12; First posted 2023-05-08 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; Diabetic neuropathy; Balance; Risk of fall; Ankle proprioceptive training
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: There will be two groups .One is interventional and the other is control group. Interventional group will be taking ankle proprioceptive training and balance training, where control will be having only balance training exercises.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participents of both groups and the outcome assessor will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iinterventional group (Experimental): Ankle proprioceptive and balance training 3 days a week for 8 weeks.
  Interventions: Other: Ankle proprioceptive training (APT); Other: Balance training (BT)
- control group (Active Comparator): Balance training 3 days a week for 8 weeks.
  Interventions: Other: Balance training (BT)

INTERVENTIONS:
Other: Ankle proprioceptive training (APT) — APT comprise of exercises including towel curls, uni-leg stance on foam with activity, writing alphabets on gym ball with toes, picking marbles with toes.
  BT includes tendem walk, side leg raises, sit to stand, side walk, back leg raise
  Arms: Iinterventional group
Other: Balance training (BT) — Balance training exercises comprising of side walk, tandem walk, standing on one leg, walking with alternating arm raise up to 90 degrees

SUMMARY:
Diabetes being a very prevalent condition results in various complications including neuropathy, which can impair various functional outcomes in patients including balance. Ankle proprioceptive training (APT) is an intervention that is used to tackle this problem. The study will compare APT with standard balance training in subjects with diabetic neuropathy.

DETAILED DESCRIPTION:
The study will include the diagnosed diabetic subjects with score of 4 or more on Douleur neuropathique 4 questionnaire (DN4Q). The subjects will be randomly divided into 2 groups; interventional group and control group. Interventional group will receive APT 3 days a week for 8 weeks. Balance training exercises will be given to both groups 3 days a week for 8 weeks. The assessments will be done at baseline, after 4 weeks and after 8 weeks of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Known case of diabetic peripheral neuropathy (DPN),
* Patients who met the criteria of DN4 scored equal or greater than 4.
* Patients who have positive SHARPEND ROMBERG TEST

Exclusion Criteria:

* Patients with DVT
* orthostatic hypotension
* Any recent surgery of lower limb
* Amputies
* Patients with crutches or walking aids
* Patients with gangrene
* Lower BMI
* Acute systemic illness
* Vestibular impairment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Mini BESTest | Baseline
  Mini BESTest is a 27-item physical performance test that distributes the items among the six sub-systems of static and dynamic balance, including stability limits/verticality, biomechanical constraints, anticipatory postural adjustments, postural responses, sensory orientation and stability in gait.
Mini BESTest | At 4 weeks
  Mini BESTest is a 27-item physical performance test that distributes the items among the six sub-systems of static and dynamic balance, including stability limits/verticality, biomechanical constraints, anticipatory postural adjustments, postural responses, sensory orientation and stability in gait.
Mini BESTest | At 8 weeks
  Mini BESTest is a 27-item physical performance test that distributes the items among the six sub-systems of static and dynamic balance, including stability limits/verticality, biomechanical constraints, anticipatory postural adjustments, postural responses, sensory orientation and stability in gait.
Sharpened Romberg (SR) | Baseline
  The Sharpened Romberg (SR) has been proposed as a quick screening tool for balance. SR requires the client to stand in tandem, with the heel of one foot touching the toe of the other foot, for 30 or 60 seconds.
Sharpened Romberg (SR) | At 4 weeks
  The Sharpened Romberg (SR) has been proposed as a quick screening tool for balance. SR requires the client to stand in tandem, with the heel of one foot touching the toe of the other foot, for 30 or 60 seconds.
Sharpened Romberg (SR) | At 8 weeks
  The Sharpened Romberg (SR) has been proposed as a quick screening tool for balance. SR requires the client to stand in tandem, with the heel of one foot touching the toe of the other foot, for 30 or 60 seconds.
Douleur Neuropathique 4 (DN4) Questionnaire | Baseline
  The Douleur Neuropathique 4 (DN4) Questionnaire is a screening tool for neuropathic pain that includes physical exams and 10 interview questions (DN4-interview). As referred in its original version scores lower than 4 were defined negative and 4 or more as positive.
Douleur Neuropathique en 4 (DN4) Questionnaire | At 4 weeks
  The Douleur Neuropathique 4 (DN4) Questionnaire is a screening tool for neuropathic pain that includes physical exams and 10 interview questions (DN4-interview). As referred in its original version scores lower than 4 were defined negative and 4 or more as positive.
Douleur Neuropathique en 4 (DN4) Questionnaire | At 8 weeks
  The Douleur Neuropathique 4 (DN4) Questionnaire is a screening tool for neuropathic pain that includes physical exams and 10 interview questions (DN4-interview). As referred in its original version scores lower than 4 were defined negative and 4 or more as positive.
Unilateral stance test | Baseline
  Unilateral stance test is used for postural stability. The participant must stand unsupported on one leg. Participants are more likely to fall hurt if they can't maintain the one-leg position for at least five seconds.
Unilateral stance test | At 4 weeks
  Unilateral stance test is used for postural stability. The participant must stand unsupported on one leg. Participants are more likely to fall hurt if they can't maintain the one-leg position for at least five seconds.
Unilateral stance test | At 8 weeks
  Unilateral stance test is used for postural stability. The participant must stand unsupported on one leg. Participants are more likely to fall hurt if they can't maintain the one-leg position for at least five seconds.
The Falls Efficacy Scale International (FES-I) | Baseline
  The Falls Efficacy Scale International (FES-I) measures people's fear about falling. FES-I scores ranging from minimum 7 (no concern about falling) to maximum 28 could be used as a rapid screening tool to evaluate a person's self-reported fear of falling.
The Falls Efficacy Scale International (FES-I) | At 4 weeks
  The Falls Efficacy Scale International (FES-I) measures people's fear about falling. FES-I scores ranging from minimum 7 (no concern about falling) to maximum 28 could be used as a rapid screening tool to evaluate a person's self-reported fear of falling.
The Falls Efficacy Scale International (FES-I) | At 8 weeks
  The Falls Efficacy Scale International (FES-I) measures people's fear about falling. FES-I scores ranging from minimum 7 (no concern about falling) to maximum 28 could be used as a rapid screening tool to evaluate a person's self-reported fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Khushnood, MSNMPT, Study Chair — Riphah International University
Locations (1):
- Capital developmental authority hospital, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No